CLINICAL TRIAL: NCT04484909
Title: Phase I Study of NBTXR3 Activated by Radiotherapy for Locally Advanced or Borderline Resectable Pancreatic Ductal Adenocarcinoma
Brief Title: NBTXR3 Activated by Radiation Therapy for the Treatment of Locally Advanced or Borderline-Resectable Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1001; NCI-2020-03731 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1001 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-06-10; First posted 2020-07-24 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Borderline Resectable Pancreatic Adenocarcinoma; Locally Advanced Pancreatic Ductal Adenocarcinoma; Resectable Pancreatic Ductal Adenocarcinoma; Stage III Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (NBTXR3, radiation therapy) (Experimental): Patients receive NBTXR3 IT on day 1. Patients then undergo 15 fractions of radiation therapy between days 15-43 in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Hafnium Oxide-containing Nanoparticles NBTXR3; Radiation: Radiation Therapy

INTERVENTIONS:
Other: Hafnium Oxide-containing Nanoparticles NBTXR3 — Given IT
  Other Names: NBTXR3
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
To find the recommended dose of NBTXR3 that can be given in combination with radiation therapy to patients with pancreatic cancer. To learn if the dose NBTXR3 found in Part 1 can help to control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

• To determine the recommended phase II dose (RP2D) of NBTXR3 activated by radiotherapy in subjects with locally advanced or borderline-resectable pancreatic ductal adenocarcinoma.

SECONDARY OBJECTIVES:

* To evaluate the safety and feasibility of NBTXR3 intratumoral injection activated by radiotherapy in locally advanced or borderline-resectable pancreatic ductal adenocarcinoma
* To evaluate the anti-tumor response of NBTXR3 intratumoral injection activated by radiotherapy in subjects with locally advanced or borderline-resectable pancreatic ductal adenocarcinoma
* To evaluate time-to-event outcomes in subjects with locally advanced or borderline-resectable pancreatic ductal adenocarcinoma

EXPLORATORY OBJECTIVES:

* To evaluate the body kinetic profile of intratumorally injected NBTXR3.
* To evaluate time to event outcomes for subjects with clinical staging of locally advanced, unresectable disease.
* To evaluate resectability conversion rates.
* To evaluate surgical outcomes in subjects who undergo surgery after radiation therapy.
* To associate radiomic measurements with outcomes.
* To evaluate biomarkers of response in subjects treated with NBTXR3/RT.

OUTLINE: This is a dose-escalation study of NBTXR3.

Patients receive NBTXR3 intratumorally (IT) on day 1. Patients then undergo 15 fractions of intensity modulated radiation therapy (IMRT) between days 15-43 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1 month and then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form (ICF) indicating that participant understands the purpose of, and procedures required for, the study and is willing to participate in the study 2. Age ≥ 18 years 3. Biopsy proven ductal adenocarcinoma of the pancreas,as defined by the following:

a. Borderline resectable pancreatic adenocarcinoma (BRPC) has no aortic involvement with at least ONE of the following features: i. Superior mesenteric vein (SMV) or Portal vein (PV) with a tumor interface of ≥ 180° OR short segment occlusion of SMV or PV amenable to reconstruction ii. Superior mesenteric artery (SMA) or celiac axis (CA) with a tumor interface of < 180° iii. Any degree of hepatic artery interface that is amenable to reconstruction b. Locally advanced pancreatic adenocarcinoma (LAPC) has at least ONE of the following features:

1. Signed informed consent form (ICF) indicating that participant understands the purpose of, and procedures required for, the study and is willing to participate in the study
2. Age ≥ 18 years
3. Biopsy proven ductal adenocarcinoma of the pancreas,as defined by the following:

   a. Borderline resectable pancreatic adenocarcinoma (BRPC) has no aortic involvement with at least ONE of the following features: i. Superior mesenteric vein (SMV) or Portal vein (PV) with a tumor interface of ≥ 180° OR short segment occlusion of SMV or PV amenable to reconstruction ii. Superior mesenteric artery (SMA) or celiac axis (CA) with a tumor interface of < 180° iii. Any degree of hepatic artery interface that is amenable to reconstruction b. Locally advanced pancreatic adenocarcinoma (LAPC) has at least ONE of the following features: i. Occlusion of the SMV or PV that is not amenable to reconstruction ii. Tumor interface of the superior mesenteric artery or celiac axis ≥ 180° iii. Involvement of the hepatic artery that is not amenable to reconstruction iv. Involvement of the aorta
4. Has had a 4-month course (± 2-months) of chemotherapy for PDAC without radiographic evidence of distant metastatic disease. Following chemotherapy regimens are allowed:

   1. gemcitabine/nab-paclitaxel
   2. gemcitabine/capecitabine
   3. gemcitabine/cisplatin
   4. gemcitabine
   5. FOLFOX
   6. FOLFIRINOX
5. Amenable to undergo the endoscopic ultrasound guided injection of NBTXR3 as per investigator or treating physician.
6. Has a target lesion in the pancreas that is identifiable on cross sectional imaging by repeated measurements (via RECIST 1.1) at the same anatomical location

   a. Nodal disease only is not allowed.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
8. Laboratory Values at screening:

   1. Hemoglobin ≥ 8.0 g/dL
   2. Absolute Neutrophil Count (ANC) ≥ 1,500/mm3
   3. Platelet Count ≥ 100,000/mm3
   4. Creatinine ≤ 1.5 x upper limit of normal (ULN)
   5. Total Bilirubin ≤ 2.0 mg/dL
   6. AST / ALT ≤ 3.0 x upper limit of normal (ULN)
   7. Serum albumin ≥ 3.0 g/dL
9. Negative pregnancy test ≤ 7 days prior to NBTXR3 injection in all females of child-bearing potential
10. If participant has a history of prior duodenal or biliar plastic stent, it should be replaced with a metal stent ≥ 1 week prior to Study Day 1.

Exclusion Criteria:

1. Prior radiation therapy to the upper abdomen
2. Prior surgical resection of pancreatic tumor
3. Diagnosis other than pancreatic ductal adenocarcinoma. All other histologic types (i.e., adenosquamous, cystadenocarcinoma, etc.) are not eligible to participate on this study.
4. LAPC or BRPC with radiographic evidence of distant metastasis at screening.
5. Has received any approved or investigational anti-neoplastic agent other than the chemotherapies specified in this protocol (i.e. chemotherapies included in Inclusion #4)
6. Known uncontrolled (Grade ≥ 2) or active gastric or duodenal ulcer disease within 30 days of enrollment
7. Known contraindication to iodine-based or gadolinium-based IV contrast
8. Active malignancy, in addition to pancreatic cancer, with the exception of basal cell carcinoma of the skin definitively treated and relapse free within at least 1 year from diagnosis
9. Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes, second or third degree atrioventricular heart block without a permanent pacemaker in place)
10. Class III or IV Congestive Heart Failure as defined by the New York Heart Association functional classification system <6 months prior to screening
11. Known active, uncontrolled (high viral load) HIV or hepatitis B or hepatitis C infection

    a. Patients who have been vaccinated for hepatitis B and do not have a history of infection are eligible.
12. Female patients who are pregnant or breastfeeding
13. Women of child-bearing potential and their male partners who are unwilling or unable to use an acceptable method of birth control for the entire study period. Acceptable methods of contraception are those that, alone or in combination, result in a failure rate of < 1% per year when used consistently and correctly
14. Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities | 4 weeks after last radiation dose
  Any grade >= 3 adverse event related to NBTXR3 and/or radiation therapy. Any toxicity (grade >= 3) that is at least possibly related to study drug (NBTXR3) is a DLT. Adverse events will be scored based on National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE v 5.0).
Maximum tolerated dose (MTD) | Up to 1 year
  MTD will be determined as the dose for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate 30%.
Recommended phase II dose (RP2D) | Up to 1 year

SECONDARY OUTCOMES:
Determination of the feasibility of NBTXR3 injection in pancreas | Up to 1 year
  Feasibility refers to the ability to do intratumoral injection of NBTXR3. The outcome for each patient would be "feasible" or "not feasible."
Progression free survival (PFS) | From NBTXR3 injection to local recurrence, local progression, distant progression, or death from any cause, whichever occurs first, assessed up to 1 year
Overall survival (OS) | From NBTXR3 injection to death from any cause or EoS, whichever occurs first, assessed up to 1 year

OTHER OUTCOMES:
Presence of hafnium | Up to 1 year
  Will evaluation of the time-course dependent presence of hafnium in blood and urine following NBTXR3 intratumoral injection.
Disease control rate | 6 months
  Defined as the proportion of patients without progression 6 months post NBTXR3 injection.
Proportion of locally advanced subjects who undergo surgical resection after receiving NBTXR3/radiation therapy (R3/RT) | Up to 1 year
Resection status | Up to 1 year
  Resection status as assessed macroscopically by surgeon R0- Macroscopically complete tumor removal with negative microscopic surgical margins, R1- Macroscopically complete tumor removal with positive microscopic margins (any or all), and R2- Macroscopically incomplete tumor removal with known or suspected residual gross disease.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene J Koay, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT04484909/ICF_000.pdf